CLINICAL TRIAL: NCT05468697
Title: A Multicenter, Open-label, Randomized, Phase 1/2 Study of Belzutifan in Combination With Palbociclib Versus Belzutifan Monotherapy in Participants With Advanced Renal Cell Carcinoma
Brief Title: A Study of Belzutifan (MK-6482) in Combination With Palbociclib Versus Belzutifan Monotherapy in Participants With Advanced Renal Cell Carcinoma (MK-6482-024/LITESPARK-024)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6482-024; MK-6482-024 (Other: MSD); LITESPARK-024 (Other: MSD); 2023-504963-17-00 (Registry Identifier: EU CT); U1111-1290-4845 (Registry Identifier: UTN)
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Renal Cell Carcinoma
Keywords: Programmed cell death ligand 1 (PD-L1); Hypoxia inducible factor 2 alpha (HIF-2 alpha); Hypoxia inducible factor 2α (HIF-2α); Renal Cell Carcinoma (RCC); Kidney Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — belzutifan; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Beltuzifan 120 mg + Palbociclib 75 mg (Experimental): Participants receive beltuzifan 120 mg orally once per day (QD) and palbociclib 75 mg orally QD in a 28-day schedule (21 days on followed by 7 days off), until progressive disease or discontinuation.
  Interventions: Drug: Belzutifan; Drug: Palbociclib
- Beltuzifan 120 mg + Palbociclib 100 mg (Experimental): Participants receive beltuzifan 120 mg orally QD and palbociclib 100 mg orally QD in a 28-day schedule (21 days on followed by 7 days off), until progressive disease or discontinuation.
  Interventions: Drug: Belzutifan; Drug: Palbociclib
- Beltuzifan 120 mg + Palbociclib 125 mg (Experimental): Participants receive beltuzifan 120 mg orally QD and palbociclib 125 mg orally QD in a 28-day schedule (21 days on followed by 7 days off), until progressive disease or discontinuation.
  Interventions: Drug: Belzutifan; Drug: Palbociclib

INTERVENTIONS:
Drug: Belzutifan — 40 mg tablet administered orally at a dose of 120 mg.
  Other Names: WELIREG™; MK-6482; PT2977
Drug: Palbociclib — 75, 100, or 125 mg tablet administered orally according to randomized dose for 21 days consecutive days followed by 7 days off.
  Other Names: IBRANCE®; PD 0332991

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of belzutifan monotherapy and belzutifan plus palbociclib combination therapy in participants with advanced clear-cell renal cell carcinoma (ccRCC) who experienced disease progression on or after receiving prior therapy. The study will establish the safety of belzutifan plus palbociclib and determine a recommended dosage of palbociclib for the combination therapy by ascending dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically confirmed diagnosis of unresectable Stage IV (per American Joint Committee on Cancer [AJCC], 8th Edition) RCC with clear-cell component
* Has had disease progression on or after having received at least 2 systemic treatments for unresectable Stage IV RCC with prior anti-programmed cell death 1 ligand 1 (PD-1/L1) and a vascular endothelial growth factor-tyrosine kinase inhibitor (VEGF-TKI) in sequence or in combination
* Has measurable disease per RECIST 1.1 as assessed by the investigator and verified by blinded independent central review (BICR)
* Has recovered from all AEs due to previous therapies

Exclusion Criteria:

* Has hypoxia, requires intermittent supplemental oxygen, or requires chronic supplemental oxygen
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has clinically significant cardiac disease
* Has moderate to severe hepatic impairment
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a history of hepatitis B (HBV) or known active hepatitis C (HCV) infection
* Has received prior treatment of belzutifan or palbociclib
* Has received prior radiotherapy ≤2 weeks prior to first dose of study intervention. Participants must have recovered from all radiation-related toxicities and not require corticosteroids
* Has had major surgery ≤3 weeks prior to first dose of study intervention
* Has received colony-stimulating factors (eg, granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM-CSF], or recombinant erythropoietin [EPO]) ≤28 days prior to the first dose of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2026-07-21 (Estimated); Study Completion 2026-07-21 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience at Least One Dose-limiting Toxicity (DLT) | Up to approximately 28 days
  A DLT consists of one or more of the following toxicities: Grade (Gr) 3 or 4 hypoxia or dyspnea; Gr 3 or 4 nausea, vomiting, or diarrhea if persistent for >48 hours despite therapy; Gr 3 or 4 cardiovascular, vascular, or thrombotic events; Nonhematologic AE ≥Gr 3 in severity with exceptions; Gr 3 rash that does not resolve within 2 weeks; Gr 3 nonhematologic toxicity if persisting despite optimal medical treatment; Gr 3 or 4 hematologic toxicities; Gr 3 or 4 febrile neutropenia; Gr 3 or 4 nonhematologic laboratory value; Any aspartate aminotransferase or alanine aminotransferase >8x the upper limit of normal (ULN) or 5 to 8x ULN persisting for >2 weeks; >2 weeks delay in dosing due to intervention-related toxicity; Intervention-related toxicity causing intervention discontinuation in the first 28 days of dosing; Missing >20% of intervention doses due to drug-related AEs; Gr 5 toxicity. The number of participants who experience at least one DLT will be reported.
Number of Participants Who Experience at Least One Adverse Event (AE) | Up to approximately 4 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience at least one AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 4 years
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. The number of participants who discontinued from the study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (13):
- United States (4):
  - Georgetown University Medical Center ( Site 1002), Washington D.C., District of Columbia
  - University of Chicago Medical Center ( Site 1007), Chicago, Illinois
  - Beth Israel Deaconess Medical Center-Cancer Clinical Trials Office ( Site 1001), Boston, Massachusetts
  - Huntsman Cancer Institute-HCI Clinical Trials Office ( Site 1004), Salt Lake City, Utah
- Australia (4):
  - Macquarie University-MQ Health Clinical Trials Unit ( Site 2001), Macquarie University, New South Wales
  - Westmead Hospital ( Site 2006), Westmead, New South Wales
  - Frankston Hospital-Oncology and Haematology ( Site 2005), Frankston, Victoria
  - One Clinical Research ( Site 2008), Nedlands, Western Australia
- Israel (5):
  - Emek Medical Center-oncology ( Site 3003), Afula
  - Rambam Health Care Campus-Oncology ( Site 3000), Haifa
  - Shaare Zedek Medical Center-Oncology ( Site 3002), Jerusalem
  - Rabin Medical Center-Oncology ( Site 3004), Petah Tikva
  - Sourasky Medical Center ( Site 3005), Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Meiman D, Skaar TC, Shugg T, Quinney SK. Physiologically Based Pharmacokinetic Model to Assess the Drug-Drug-Gene Interaction Potential of Belzutifan in Combination With Cyclin-Dependent Kinase 4/6 Inhibitors. JCO Precis Oncol. 2025 Jul;9:e2500153. doi: 10.1200/PO-25-00153. Epub 2025 Jul 25. PMID 40712111
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26125&tenant=MT_MSD_9011